CLINICAL TRIAL: NCT02275377
Title: Effects of Inspiratory Muscle Training on Blood Pressure Levels in Hypertensive Individuals: a Randomized Clinical Trial.
Brief Title: Effects of Inspiratory Muscle Training on Blood Pressure Levels in Hypertensive Individuals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 14-0405
Record Dates: First submitted 2014-09-30; First posted 2014-10-27 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Hypertension
Keywords: Breathing Exercises; Autonomic Control; Blood Pressure.
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Inspiratory muscle training (IMT) (Experimental): Participants will be submitted to a linear pressure resistance (PowerBreathe) with an inspiratory load of 40% of maximal inspiratory pressure (adjusted weekly), seven days a week, session duration of 30 minutes for 8 weeks.
  Interventions: Other: Inspiratory muscle training (IMT)
- Sham IMT (Placebo Comparator): Participants will be submitted to inspiratory muscle training with the same equipment as the intervention group, but without a load generating resistance.
  Interventions: Other: Sham IMT
- Normotensive (No Intervention): The normotensive control group (healthy) will go through the same initial evaluation without performing inspiratory muscle training.

INTERVENTIONS:
Other: Inspiratory muscle training (IMT) — Participants will receive IMT for 30 min, 7 times per week for 8 weeks using Inspiratory muscle trainer device (PowerBreathe). During training, participants will be instructed to maintain diaphragmatic breathing with a breathing rate of 15-20 cycles/min. Inspiratory load will be set at 40% of maximum static inspiratory pressure, and weekly training loads will be adjusted to maintain 40% of MIP. Each week, six training sessions will be held at home and a training session will be supervised in the research center.
  Other Names: Inspiratory muscle training
  Arms: Inspiratory muscle training (IMT)
Other: Sham IMT — Participants will receive IMT for 30 min, 7 times per week for 8 weeks using Inspiratory muscle trainer device (PowerBreathe). During training, participants will be instructed to maintain diaphragmatic breathing with a breathing rate of 15-20 cycles/min, but without a load generating resistance. Each week, six training sessions will be held at home and a training session will be supervised in the research center.
  Other Names: Sham Inspiratory muscle training
  Arms: Sham IMT

SUMMARY:
This research aims to evaluate the effects of inspiratory muscle training (IMT) on blood pressure, in inspiratory muscle mechanoreflex, autonomic cardiovascular control in subjects with hypertension.

DETAILED DESCRIPTION:
Patients with hypertension will be selected through the Outpatient Hypertension of the Hospital of Clinics de Porto Alegre, for convenience. Subsequently, patients will be subjected to test respiratory muscle strength (manometer), respiratory muscle resistance, cardiopulmonary exercise testing (maximum), evaluation of cardiac reflex sensitivity and autonomic control test and induction of inspiratory muscle mechanoreflex with occlusion plethysmography at baseline before the start of the training protocol. Patients will randomize inspiratory muscle training for 30 minutes a day, 7 days a week, for 8 weeks with muscle training device (PowerBreathe). There will be a weekly monitoring in the Clinical Research Center of the institution where the maximal inspiratory pressure (MIP) and respiratory training techniques will be reassessed and readjusted (40% of MIP). The control group will be submitted to respiratory training techniques with muscle training device (PowerBreathe) without load. After this period, all initial tests will be reassessed. A healthy control group study with 10 normotensive individuals will be included.

ELIGIBILITY:
Inclusion Criteria:

Participants will be selected from the medical records in search of Basic Health Unit and Hypertension Clinic - Hospital of Clinics of Porto Alegre (HCPA), Porto Alegre - RS:

* Diagnosis of essential hypertension with systolic blood pressure ≥140 mmHg and / or diastolic blood pressure ≥ 90 mmHg without treatment or use of antihypertensive;
* Only taking diuretics (monotherapy) or none;
* Body mass index ≤ 29.9 kg / m²;
* Not engaged in physical activity;
* Inspiratory muscle strength ≥ 70% of predicted.

  * Inclusion of normotensive individuals with systolic blood pressure <130 mmHg and/or diastolic blood pressure <85 mmHg by ambulatory blood pressure monitoring (ABPM).

Exclusion Criteria:

* Blood pressure ≥ 160/100 mmHg
* Pregnant and lactating women;
* Deep vein thrombosis; current or previous.
* Diabetes mellitus;
* Orthopedic impairments, musculoskeletal, neurological and / or cognitive impairment, or even other diseases that compromise participation in the proposed protocol;
* Acute myocardial infarction within the last 6 months;
* Hearth failure;
* Angina pectoris;
* Pulmonary impairment from any source;
* Current smoking.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-10 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Levels of blood pressure (mmHg) | 8 weeks
  Ambulatory blood pressure monitoring (ABPM).

SECONDARY OUTCOMES:
Inspiratory muscle mechanoreflex | 8 weeks
  Venous occlusion plethysmography measure during inspiratory muscle training exercise at 60% and 2% of maximal inspiratory muscle strength.
Cardiopulmonary Capacity | 8 weeks
  High-intensity exercise test (maximum) assessed by ergometry with noninvasive hemodynamic monitoring (electrocardiogram, exhaled gas analyzer, heart rate, respiratory rate and blood pressure).
Autonomic cardiovascular control | 8 weeks
  Heart rate and blood pressure monitoring in the time domain (spectral analysis).

CONTACTS AND LOCATIONS:
Overall Officials: Leila B Moreira, PhD, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Leila Moreira, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Posser SR, Callegaro CC, Beltrami-Moreira M, Moreira LB. Effect of inspiratory muscle training with load compared with sham training on blood pressure in individuals with hypertension: study protocol of a double-blind randomized clinical trial. Trials. 2016 Aug 2;17:382. doi: 10.1186/s13063-016-1514-y. PMID 27484507